CLINICAL TRIAL: NCT01911221
Title: A Phase 3b, Single-Center, Open-label Study to Assess the Immunogenicity and Safety of Novartis Meningococcal B Recombinant Vaccine When Administered at a 0, 2-Month Schedule in Healthy At-Risk Adults Aged 18 to 65 Years Inclusive.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V72_59; 2012-005815-25 (EudraCT Number)
Record Dates: First submitted 2013-07-26; First posted 2013-07-30 (Estimated); Results first posted 2014-10-31 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Prevention of the Meningococcal Disease
Keywords: Meningococcal disease,; Adults
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rMenB+OMV NZ (Experimental): A single 0.5mL dose of the study vaccine will be administered intramuscularly in the deltoid muscle.
  Interventions: Biological: rMenB+OMV NZ

INTERVENTIONS:
Biological: rMenB+OMV NZ — Recombinant MenB with Outer Member Vesicle (OMV) from the New Zealand strain

SUMMARY:
The study will evaluate the immunogenicity and safety of the rMenB+OMV NZ in an adult population potentially at risk for meningococcal disease (e.g. lab workers).

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 65 years of age inclusive who have given written informed consent at the time of enrollment;
2. Who are available for all the visits scheduled in the study (i.e., not planning to leave the area before the end of the study period);
3. In good health as determined by medical history, physical examination and clinical judgment of the investigator;
4. Who are or might be routinely exposed to cultures of N. meningitidis serogroup B.

Sponsor's employees are considered eligible to participate in the trial as per inclusion criteria.

Exclusion Criteria:

1. Pregnancy or nursing (breastfeeding) mothers;
2. Females of reproductive age who have not used or do not plan to use acceptable birth control measures, for the 3 months duration of the study. Oral, injected or implanted hormonal contraceptive, diaphragm, condom, intrauterine device or sexual abstinence are considered acceptable forms of birth control. If sexually active the subject must have been using one of the accepted birth control methods for at least 60 days prior to study entry;
3. Any serious chronic or progressive disease according to judgment of the investigator (e.g. neoplasm, insulin dependent diabetes, cardiac, renal or hepatic disease);
4. Individuals with history of any progressive or severe neurologic disorder, or seizure disorder. A single episode of febrile convulsion is not an exclusion criteria;
5. History of any serogroup B meningococcal vaccine administration;
6. Previous known or suspected disease caused by N. meningitidis;
7. History of severe allergic reaction after previous vaccinations, or hypersensitivity to any component of the vaccine;
8. Known or suspected autoimmune disease or impairment/alteration of the immune system resulting from (for example):

   * Receipt of any chronic immunosuppressive therapy
   * Receipt of any chronic immunostimulants
   * Immune deficiency disorder, or known HIV infection
9. Subjects who are not able to comprehend and to follow all required study procedures for the whole period of the study;
10. History or any illness/condition that, in the opinion of the investigator, might interfere with the results of the study or pose additional risk to the subjects due to participation in the study;
11. Any significant chronic infection;
12. Known bleeding diathesis or any condition that may be associated with a prolonged bleeding time;
13. Family members and household members of research staff;
14. Participation in another clinical trial within the last 30 days or planned for during study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (1):
- Novartis site, Marburg, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from single study center in Germany.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- rMenB+OMV NZ: Subjects received two doses of rMenB +OMV NZ at 0 month and 2 month schedule.
Period: Overall Study
Arm/Group | rMenB+OMV NZ
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Subjects received two doses of rMenB+OMV NZ at 0 month and 2 month schedule.
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: year] | 38.5 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 10
  MALE | 3

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Human Serum Bactericidal Activity Titers Against N Meningitidis Serogroup B Strains Following A Two-dose Vaccination Schedule
Description: The immunogenicity was assessed to evaluate the human serum bactericidal activity (hSBA) against the indicator strains of N meningitidis serogroup B (H44/76, 5/99, NZ98/254) and M10713 strain at baseline and at one month after the second vaccination.
Time Frame: Day1 and Day 91
Population: Analysis was done on Full Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Groups:
- rMenB+OMV NZ: Subjects received two doses of rMenB +OMV NZ vaccine at 0 and 2 month schedule.
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 13
Titers
  H44/76 Prevaccination (Day 1) | 1.18 [0.92 to 1.52]
  Post 2nd vaccination (Day 91) | 53 [34 to 84]
  5/99 Prevaccination (Day 1) | 2.27 [1.34 to 3.85]
  After 2nd vaccination (Day 91)(N=12) | 143 [57 to 356]
  NZ98/254 Prevaccination (Day 1) | 1.09 [0.91 to 1.31]
  Post 2nd vaccination (Day 91)(N=12) | 15 [5.41 to 43]
  M10713 Prevaccination (Day 1) | 21 [12 to 39]
  Post second vaccination (Day 91)(N=12) | 56 [31 to 99]

2. Primary Outcome: Geometric Mean Ratios Against N Meningitidis Serogroup B Strains Following A Two-dose Vaccination Schedule
Description: The immunogenicity was assessed to evaluate the hSBA in terms of geometric mean ratios within subjects against the indicator strains of N meningitidis serogroup B (H44/76, 5/99, NZ98/254) and strain M10713 at one month after the second vaccination versus baseline.
Time Frame: Day1 and Day 91
Population: The analysis was done on the Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 13
ratio
  H44/76 (Day 91/Day 1) | 45 [29 to 70]
  5/99 (Day 91/Day 1)(N=12) | 59 [21 to 166]
  NZ98/254 (Day 91/Day 1)(N=12) | 14 [5.17 to 37]
  M10713 (Day 91/Day 1)(N=12) | 2.99 [1.43 to 6.27]

3. Primary Outcome: Percentages Of Subjects With hSBA≥ 1:5 Titers Against N Meningitidis Serogroup B Strains Following Two-Dose Vaccination Schedule.
Description: The immunogenicity was assessed to evaluate the hSBA titers ≥ 1:5 in terms of percentages of subjects against N meningitidis serogroup B (H44/76, 5/99, NZ98/254) and strain M10713 following a two dose vaccination schedule with rMenB+OMV NZ vaccine.
Time Frame: Day1 and Day91
Population: Analysis was done on Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 13
Percentages of subjects
  H44/76 Prevaccination (Day 1) | 0 [0 to 25]
  Post 2nd vaccination (Day 91) | 100 [75 to 100]
  5/99 Prevaccination (Day 1) | 31 [9 to 61]
  After 2nd vaccination (Day 91)(N=12) | 100 [74 to 100]
  NZ98/254 Prevaccination (Day 1) | 0 [0 to 25]
  Post 2nd vaccination (Day 91)(N=12) | 75 [43 to 95]
  M10713 Prevaccination (Day 1) | 92 [64 to 100]
  Post second vaccination (Day 91)(N=12) | 100 [74 to 100]

4. Primary Outcome: Percentages Of Subjects With hSBA≥ 1:8 Titers Against N Meningitidis Serogroup B Strains Following Two-Dose Vaccination Schedule.
Description: The immunogenicity was assessed to evaluate the human serum bactericidal activity titers ≥ 1:8 in terms of percentages of subjects against N meningitidis serogroup B (H44/76, 5/99, NZ98/254) and strain M10713 following a two dose vaccination schedule with rMenB+OMV NZ vaccine.
Time Frame: Day1 and Day91
Population: Analysis was done on Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 13
Percentage of Subjects
  H44/76 Prevaccination (Day 1) | 0 [0 to 25]
  Post 2nd vaccination (Day 91) | 100 [75 to 100]
  5/99 Prevaccination (Day 1) | 8 [0 to 36]
  After 2nd vaccination (Day 91)(N=12) | 92 [62 to 100]
  NZ98/254 Prevaccination (Day 1) | 0 [0 to 25]
  Post 2nd vaccination (Day 91)(N=12) | 75 [43 to 95]
  M10713 Prevaccination (Day 1) | 85 [55 to 98]
  Post second vaccination (Day 91)(N=12) | 92 [62 to 100]

5. Primary Outcome: Percentages Of Subjects With Four-Fold Increase In Human Serum Bactericidal Activity From Baseline Against N Meningitidis Serogroup B Strains Following a Two Dose Vaccination Schedule.
Description: The antibody responses were assessed to evaluate the four fold increase in human serum bactericidal activity titers in terms of percentages of subjects against N meningitidis serogroup B (H44/76, 5/99, NZ98/254) and strain M10713 following a two dose vaccination schedule with rMenB+OMV NZ vaccine.
Time Frame: Day 91
Population: Analysis was done on Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 13
Percentage of subjects
  H44/76 | 100 [75 to 100]
  5/99 (N=12) | 92 [62 to 100]
  NZ98/254 (N=12) | 75 [43 to 95]
  M10713 (N=12) | 33 [10 to 65]

6. Primary Outcome: Geometric Mean Concentrations For Vaccine Antigen 287-953 Following A Two-dose Vaccination Schedule
Description: The antibody responses were assessed to evaluate the geometric mean concentrations as measured by Enzyme Linked Immunosorbent Assay (ELISA) in terms of percentages of subjects for the vaccine antigen 287-953 following a two dose vaccination schedule with rMenB+OMV NZ vaccine at baseline and at one month the second vaccination.
Time Frame: Day 1 and Day 91
Population: Analysis was done on Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: U/mL
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 13
U/mL
  Prevaccination (Day 1) | 22 [18 to 28]
  Post second vaccination (Day 91) | 1200 [537 to 2680]

7. Primary Outcome: Geometric Mean Ratios For Vaccine Antigen 287-953 Following A Two-dose Vaccination Schedule.
Description: The antibody responses were assessed to evaluate the geometric mean ratios as measured by ELISA within the subjects for the vaccine antigen 287-953 following a two dose vaccination schedule with rMenB+OMV NZ vaccine at one month after the second vaccination versus baseline.
Time Frame: Day 1 and Day 91
Population: Analysis was done on Full Analysis Set.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 13
Ratio | 54 [24 to 120]

8. Primary Outcome: Percentages of Subjects With Four Fold Increase From Baseline For Vaccine Antigen 287-953 Following A Two-dose Vaccination Schedule.
Description: The antibody responses were assessed to evaluate the four fold increases in ELISA concentrations as measured by ELISA to the vaccine antigen 287-953 following a two dose vaccination schedule with rMenB+OMV NZ vaccine at one month the second vaccination over baseline.
Time Frame: Day 1 and Day 91
Population: Analysis was done on Full Analysis Set.
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 13
Percentage of Subjects | 85 [55 to 98]

9. Primary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events After Receiving rMenB+OMV NZ Vaccine ( After Any Vaccination)
Description: The number of subjects with solicited local and systemic adverse events after receiving rMenB+OMV NZ (a two dose vaccination schedule) collected from day 1 through day 7 are reported.
Time Frame: Day 1 through Day 7 postvaccination.
Population: Analysis was done on Solicited Safety Set.
Measure: Number; unit: Number of Subjects
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 13
Number of Subjects
  Any local | 13
  Injection site erythema | 0
  Injection site swelling | 0
  Injection site induration | 1
  Injection site pain | 13
  Any Systemic | 9
  Nausea | 2
  Myalgia | 3
  Arthralgia | 3
  Fatigue | 5
  Headache | 8
  Fever (≥38°C) | 1
  Prophylactic use of antipyretics/analgesics | 0
  Therapeutic use of antipyretics/analgesics | 4

10. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Receiving rMenB+OMV NZ Vaccine ( After Any Vaccination).
Description: Safety was assessed as the number of subjects who reported unsolicited adverse events as collected from Day 1 to Day 91 following rMenB+OMV vaccination (a two dose schedule). Unsolicited adverse events were collected from day 1 through day 7 after each vaccination, while serious adverse events, medically attended adverse events and adverse events leading to withdrawal from study were reported from day 1 through day 91.
Time Frame: Day 1 through Day 91 postvaccination.
Population: Analysis was done on Unsolicited Safety Set.
Measure: Number; unit: Number of subjects
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 13
Number of subjects
  Any unsolicited AEs | 8
  At least possibly related unsolicited AEs | 7

11. Primary Outcome: Number of Subjects Reporting Unsolicited Serious Adverse Events After Receiving rMenB+OMV NZ Vaccine ( After Any Vaccination).
Description: Safety was assessed as the number of subjects who reported Serious Adverse Events (SAEs), medically attended AEs, AEs leading to withdrawal from the study, as collected from day 1 to day 91 following vaccination with rMenB+OMV NZ (a two dose schedule ) are reported.
Time Frame: Day 1 through Day 91 postvaccination.
Population: Analysis was done on Unsolicited Safety Set.
Measure: Number; unit: Number of subjects
Arm/Group | rMenB+OMV NZ
Number analyzed (Participants) | 13
Number of subjects
  AEs leading to study withdrawal | 0
  Medically attended AEs | 2
  Any SAEs | 0
  At least possibly related SAEs | 0
  AEs leading to death | 0

ADVERSE EVENTS:
Time Frame: Day 1 through Day 91 postvaccination.
Description: Safety was assessed as the number of subjects who reported Serious Adverse Events (SAEs), medically attended AEs, AEs leading to withdrawal from the study, as collected from day 1 to day 91 following vaccination with rMenB+OMV NZ (a two dose schedule ) are reported.
Groups:
- rMenB+OMVNZ: Subjects received two doses of rMenB +OMV NZ at 0 month and 2 month schedule.
Arm/Group | rMenB+OMVNZ
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 13/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rMenB+OMVNZ (N=13)
NAUSEA (Gastrointestinal disorders) | 2
CHILLS (General disorders) | 1
FATIGUE (General disorders) | 5
INJECTION SITE ERYTHEMA (General disorders) | 10
INJECTION SITE INDURATION (General disorders) | 5
INJECTION SITE PAIN (General disorders) | 13
INJECTION SITE SWELLING (General disorders) | 5
PYREXIA (General disorders) | 1
NASOPHARYNGITIS (Infections and infestations) | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3
MYALGIA (Musculoskeletal and connective tissue disorders) | 3
HEADACHE (Nervous system disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days